CLINICAL TRIAL: NCT02989545
Title: The Use of an "Anal-Tape" in Patients With Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dan Livovsky, Dr. Dan M. Livovsky and Dr. Joseph Lysy, Shaare Zedek Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Shaare Zedek Medical Center FI
Record Dates: First submitted 2016-12-07; First posted 2016-12-12 (Estimated); Results first posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Off treatment (No Intervention): 2 week period without intervention
- Treatment period (Experimental): 2 week period with intervention
  Interventions: Device: Anal Tape

INTERVENTIONS:
Device: Anal Tape
  Arms: Treatment period

SUMMARY:
Fecal incontinence (FI), defined as the involuntary passage of stool for more than 3 months and is a devastating disease. The negative impact on quality of life has been consistently demonstrated. The prevalence of FI is probably underestimated in most studies. Currently conservative treatment is only modestly effective and surgical treatment is complex and expensive with less than optimal efficacy.

The investigators developed an "anal tape" using a commercially available elastic band with a special adhesive that is approved for use in the skin. A special design of the tape can be applied to the skin surrounding the anus providing support and additional pressure forces to the anal sphincter.

This is a 4 week, prospective, non blinded, cross-over study to explore the efficacy and safety of this device in patients with FI. The primary endpoint will be improvement in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Fecal incontinence for more than 6 months
* Willing to participate
* Understand the study procedures
* Is able to apply and remove the "anal tape" without significant assistance of others.
* Have done sigmoidsocopy or colonoscopy and anal manometry within five year of screening visit

Exclusion Criteria:

* Advanced full thickness rectal prolapse.
* Injured, inflamed or any significant disease in the peri-anal skin.
* Allergy to any component of the device, either known or developed during testing in the screening visit.
* Moderate to severe proctitis of any etiology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

REFERENCES:
- [Derived] Livovsky DM, Koslowsky B, Goldin E, Lysy J. External kinesiology tape for improvement in fecal incontinence symptom bother in women: a pilot study. Int Urogynecol J. 2022 Oct;33(10):2859-2868. doi: 10.1007/s00192-021-05050-z. Epub 2022 Jan 18. PMID 35039916

RESULTS

PARTICIPANT FLOW:
Groups:
- Per Sequence: Off treatment first for 14 days Treatment period second for 14 days
Period: Control Period - no Intervention
Arm/Group | Per Sequence
Started | 20
Completed | 20
Not Completed | 0
Period: Treatment Period - Anal Tape Provided
Arm/Group | Per Sequence
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: 2 week period without intervention then 2 week period with anal tape intervention
Arm/Group | All Patients
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 64 [56.5 to 69.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 20

OUTCOME MEASURES:

1. Primary Outcome: Any Improvment in the Fecal Incontince Quality of Life Scale (FIQoLs)
Description: The FIQoL is a validated, condition-specific tool that evaluates quality of life (QoL) in patients with fecal incontinence (FI) it consisting of 29 questions, subdivided into four domains: Lifestyle, Coping/Behavior, Depression/Self-perception, and Embarrassment. Item 1, general health, is graded from 1 "excellent" to 5 "poor" and is reversely scored. Items 2 to 28 are graded on a 4-point Likert-scale (1 = lower QoL). Item 29, FI specific depression, is graded from 1 "extremely so" to 6 "not at all." The average score for each domain is calculated separately and is calculated only if half or more of the items in the particular domain have been answered. Scales range from 1 to 5, with a 1 indicating a lower quality of life. Each domain or subscale is reported separately (Range 1 to 5), a total score including all four domains is not calculated.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Treatment Period: 2 week period with intervention - Anal tape
Arm/Group | Off Treatment | Treatment Period
Number analyzed (Participants) | 20 | 20
score on a scale
  Lifestyle | 2.8 (0.69) | 3.3 (0.68)
  Coping/Behaivoir | 1.9 (0.64) | 2.5 (0.73)
  Depression/Self-Perception | 3.1 (0.75) | 3.5 (0.74)
  Embarrassment | 2.13 (0.67) | 2.65 (0.76)

2. Secondary Outcome: A 50% Reduction in the Number of Episodes of FI Per Week
Description: Number of pateints with reduction of more than 50% in the absolute number of FI events during each week of the study
Time Frame: 4 weeks
Population: Note that this outcome was obtained by free text stool diaries that patients had to keep at home. Only 15 patient out of 20 provided full diaries, therefore the analysis is limited to 15 instead of all 20.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Period: 2 week period with intervention
  Anal Tape
Arm/Group | Off Treatment | Treatment Period
Number analyzed (Participants) | 15 | 15
Participants | 0 | 5

3. Secondary Outcome: Mean Wexner Score
Description: The Wexner Scale is a measure of frequency and severity of anal incontinence. It comprises five items, three regarding frequency of involuntary passage of gas, liquid, or solid stool, frequency of pad wearing, and frequency of lifestyle alteration, scored in a 5-point Likert-scale (never=0, rarely=1, sometimes=2, usually=3, always=4). A sum of all scores from 0 to 20 is calculated with higher scores meaning more severe incontince.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Off Treatment | Treatment Period
Number analyzed (Participants) | 20 | 20
score on a scale | 11.9 (3.5) | 10.3 (4.8)

4. Secondary Outcome: Mean Redction in Wexner Scale Compared to Baseline
Description: as for outcome 3
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Off Treatment | Treatment Period
Number analyzed (Participants) | 20 | 20
score on a scale | 0.6 (1.7) | 1.95 (4.2)

5. Secondary Outcome: General Satisfaction
Description: General satisfaction with the device was assessed using a standard 100 mm visual analog scale. Patients were asked to grade their satisfaction with the device between 0 and 100 by drawing a perpendicular line in the 100 mm visual analog scale. Then the distance in mm was measured in mm from 0 to the perpendicular line and the score was calculated. Higher scores meaning better satisfaction.
Time Frame: 2 weeks
Population: Note that in 3 patients these data were missing, therefore the analysis if for 17 out of 20 participants.
Measure: Median (Inter-Quartile Range); unit: mm in VAS scale
Arm/Group | Treatment Period
Number analyzed (Participants) | 17
mm in VAS scale | 80 [50 to 90]

6. Secondary Outcome: Willingness of the Patient to Continue Using the Anal Tape After the Study.
Description: Willingness of the patient to continue using the device was assessed using a standard 100 mm visual analog scale. Patients were asked to grade their willingness to use the device in the future between 0 and 100 by drawing a perpendicular line in the 100 mm visual analog scale. Then the distance in mm was measured in mm from 0 to the perpendicular line and the score was calculated. Higher scores meaning better satisfaction.
Time Frame: 4 weeks
Population: Note that in 3 patients these data were missing, therefore the analysis if for 17 out of 20 participants.
Measure: Median (Inter-Quartile Range); unit: mm in VAS scale
Arm/Group | Treatment Period
Number analyzed (Participants) | 17
mm in VAS scale | 90 [50 to 90]

ADVERSE EVENTS:
Time Frame: 4 weeks study period
Groups:
- Control Period - No Intervention: Consiting of the first 14 days of the study during which patients were off treatment and baseline and safety data was collected
- Treatment Period - Anal Tape Provided: Consiting of the second 14 days of the study (day 15 to 28) during which patients were provided with the "anal tape" device and during this period efficacy and safety data was collected.
Arm/Group | Control Period - No Intervention | Treatment Period - Anal Tape Provided
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Period - No Intervention (N=20) | Treatment Period - Anal Tape Provided (N=20)
Mild difficulty to remove the device (Gastrointestinal disorders) | 0 (0) | 3 (3) — Mild difficulty to remove the device

LIMITATIONS AND CAVEATS:
Short term, single center, open label

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT02989545/Prot_SAP_000.pdf